CLINICAL TRIAL: NCT00733694
Title: Clinical Evaluation of the Low Contact Stress (LCS) Classic and Universal Mobile-bearing Total Knee System. The Asian LCS User Group - 'The Dragon Knee Study'
Brief Title: Outcome Study of Total Knee Arthroplasty in Asian Patients
Acronym: DRAGON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT 99/33
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: Arthroplasty, Replacement, Knee,LCS
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCS® Complete™ Mobile Bearing Knee Systems (Other): An orthopaedic implant for primary total knee replacement with a mobile bearing knee
  Interventions: Device: LCS® Complete™ Mobile Bearing Knee Systems

INTERVENTIONS:
Device: LCS® Complete™ Mobile Bearing Knee Systems — An orthopaedic implant for primary total knee replacement with a mobile bearing knee

SUMMARY:
To determine how the LCS mobile bearing knee system works within the Asian Population.

DETAILED DESCRIPTION:
The objective of this clinical evaluation is to compile a profile of the performance of the LCS Mobile bearing total knee system in normal clinical practice within the Asian Population. Performance will be assessed using specific surgeon and patient based outcome scores.

Total subject enrolled 505; 6 subjects did not receive device. Total subjects received device 499.

Among those who received devices, 391 subjects unilateral and 108 bilateral, therefore, total 607 knees in the study

ELIGIBILITY:
Inclusion Criteria:

* Administrative - the patient is able to understand the evaluation, is able to give consent and will comply with the postoperative follow up regime.
* Diagnosis - idiopathic osteoarthritis, rheumatoid arthritis, post traumatic arthritis or any other pathology that in the opinion of the clinical investigator requires a primary total knee arthroplasty.
* Implant suitability - patients who in the opinion of the Clinical Investigator are considered suitable for treatment with a mobile bearing knee system (the LCS Classic or Universal).
* Bilateral patients - simultaneous bilateral patients are included. Staged bilateral patients are included if the second procedure is performed within the one-year recruitment period. Staged bilateral patients where the second procedure is performed outside of the one-year recruitment period will only be included if the second procedure is performed within 6 months of the end of the one-year recruitment period.
* Age - the upper age limit is set at 75 years and expected to live through the 5 years study period.vi. Ethnic Origin - patients must be Asian in ethnic origin
* Unicondylar / High Tibial Osteotomy (HTO) conversion - patients that are being converted from a unicondylar / HTO procedure are included providing the reason for conversion is due to progression of the disease process affecting the other condyle. Patients that are converted and have evidence of infection / aseptic loosening / loss of bone stock are excluded.

Exclusion Criteria:

* Patients with a known history of poor compliance to medical treatment.
* Patients that require revision surgery
* Patients with gross ligamentous insufficiency.
* Patients with a severe valgus deformity (15 degrees or greater)
* Patients with a severe varus deformity (20 degrees or greater)
* Patients with a fixed flexion contracture (30 degrees or greater)
* Patients over the age of 75 years.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2000-04-01 (Actual); Primary Completion 2008-04-01 (Actual); Study Completion 2008-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Oxford Knee Score | 5 years
  Oxford Knee Score will be summarized pre-operatively and at each subsequent post-operative follow-up. The change from pre-op to final post-operative assessment at 5 years will be derived and used as the analysis variable.

SECONDARY OUTCOMES:
Change in Quality of Life Score (SF-36), Knee Society Score, Anterior Pain and radiographic/radiolucent details from pre-op to 5 year post-op follow up. | 5 years
Adverse Events | 5 years
  All intraoperative and postoperative adverse incidences/complications and their relationship to the knee will be collected

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedic Surgery University of Hong Kong, Hong Kong, China